CLINICAL TRIAL: NCT03178786
Title: Visual Spatial Exploration and Art Therapy Intervention in Patients Diagnosed With Parkinson's Disease
Acronym: ExplorArtPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-00191
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: Art Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease (Experimental)
  Interventions: Behavioral: PAT sessions
- Healthy Control Subjects (Sham Comparator)
  Interventions: Behavioral: PAT sessions

INTERVENTIONS:
Behavioral: PAT sessions — PD subjects will be tested twice, that is, within four weeks before (Baseline) and after the completion of 9 PAT projects (Follow up).

SUMMARY:
The purpose of this dual phase cross-sectional, controlled and prospective, open label, exploratory study is to determine the general characteristics of visuospatial exploration and its neural substrate in subjects with Parkinson's Disease (PD) and to explore the impact of professional art therapy intervention in a cohort of subjects with Parkinson's Disease on visuospatial exploration, visuomotor integration, neuropsychological and emotional sphere, quality of daily living and motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Patients with PD)

* Diagnosis of PD according to United Kingdom Parkinson's Disease Society Brain Bank;
* Hoehn and Yahr stage 2 to 3;

Exclusion Criteria:

Exclusion Clinical Criteria (For both PD and Controls):

* History of dementia, or MoCA < 22;
* Untreated depression, or score of >20 on Beck Depression Inventory II;
* History of florid visual, tactile, olfactory or acoustic hallucinations requiring the administration of neuroleptics.
* Presence of psychosis requiring the administration of neuroleptics or sedatives.
* Presence of severe motor fluctuations with most of the 50% of day spent in off-time.
* Presence of bothersome dyskinesias.
* Presence of severe dystonia involving the head-neck axis including anterocollis, laterocollis and torticollis.
* Presence of severe fluctuations in attention, alertness or cognition.
* Presence of any clinically significant abnormality on vital signs.

Exclusion Ophthalmologic and Ophtalmometric Criteria (For both PD and Controls):

* Visual abnormalities requiring exclusive correction with eye glasses (of note, contact lenses are NOT an exclusion criterion).
* History of clinically active ophthalmologic abnormalities including but not limited to macular degeneration, symptomatic cataract, symptomatic retinopathy, recent orbital trauma with periorbital ecchymosis, symptomatic thyroid eye disease, refractory problems of moderate or severe degree (of note, mild refractory problems are NOT an exclusion criterion, chromatic discrimination problems including daltonism are NOT an exclusion criterion).
* History of any clinically significant CNS abnormality resulting in an active visual field deficit including but not limited to brain tumors, brain abscess, inflammatory encephalic lesions, traumatic brain injury or stroke.
* Clinically significant abnormal findings on routine bedside examination of the vision system during a standard clinical neurological exam.

Exclusion MRI Criteria (For both PD and Controls):

* Major or unstable medical illness;
* Left hand dominance;
* Pacemakers, neurostimulators, intracranial clips, metal implants, external clips or metal foreign bodies within 10 cm of the head;
* Current pregnancy or nursing;
* Pregnancy planned;
* Claustrophobia;
* Large body habitus (280 lb or more)

Exclusion Criteria for Art Therapy (For PD subjects only):

* Severe inability to perform line drawing;
* Severe inability to manipulate soft/light materials like clay.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Eye Movement Analysis | 19 Weeks
  Eye positions will be recorded for both eyes concurrently. The system will record binocularly with a sampling frequency of 250Hz and a spatial accuracy of 0.5 degrees, approximately. Eye movement data will be analyzed off-line using customized MATLAB software (www.mathworks.com).
Rey-Osterrieth Complex Figure Test | 19 Weeks
  These tests explore different aspects of visuospatial abilities including attention, memory, abstraction, planning and visuoexecutive skills; neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing, first by copying it freehand (recognition), and then drawing from memory (recall)
Benton test | 19 Weeks
  These tests explore different aspects of visuospatial abilities including attention, memory, abstraction, planning and visuoexecutive skills; individually administered test for people aged from eight years to adulthood that measures visual perception and visual memory. It can also be used to help identify possible learning disabilities among other afflictions that might affect an individual's memory. The individual examined is shown 10 designs, one at a time, and asked to reproduce each one as exactly as possible on plain paper from memory.
Corsi Block Test | 19 Weeks
  These tests explore different aspects of visuospatial abilities including attention, memory, abstraction, planning and visuoexecutive skills; psychological test that assesses visuo-spatial short term working memory. It involves mimicking a researcher as he/she taps a sequence of up to nine identical spatially separated blocks.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Cucca, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States